CLINICAL TRIAL: NCT02370277
Title: Changes in Intestinal Microbiota in Association With Chemotherapy Treatment
Brief Title: Effects of Chemotherapy on Intestinal Bacteria in Patients With Newly Diagnosed Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1B-14-6; NCI-2014-02611 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-14-00712; 1B-14-6 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Ductal Breast Carcinoma In Situ; Invasive Breast Carcinoma; Stage I Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, blood, and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A (stool collection after adjuvant chemotherapy): Patients undergo collection of stool samples at baseline (before surgery), at 1 week before initiation of adjuvant chemotherapy (after surgery), and at 1 and 4 months after completion of adjuvant chemotherapy.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Group B (stool collection after adjuvant chemotherapy): Patients undergo collection of stool samples at baseline (after surgery), at 1 week before initiation of adjuvant chemotherapy, and at 1 and 4 months after completion of adjuvant chemotherapy.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Group C (stool collection after neoadjuvant chemotherapy): Patients undergo collection of stool samples at baseline, 1 month after completion of neoadjuvant chemotherapy (before surgery), and at 1 and 4 months after surgery
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of stool samples
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot research trial studies the effects of chemotherapy on intestinal bacteria/organisms (microbiota) in patients newly diagnosed with breast cancer. Change in intestinal microbiota may be associated with weight gain in patients treated with chemotherapy. Weight gain has been also associated with cancer recurrence. Examining the types and quantity of bacterial composition in the stool of breast cancer patients treated with chemotherapy may help determine whether body weight and composition are associated with changes in the intestinal microbiota and allow doctors to plan better treatment to prevent weight gain and possibly disease recurrence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the transitory and longer lasting effects of chemotherapy on the gut microbiota.

SECONDARY OBJECTIVES:

I. To examine the relationship between body composition and gut microbiota before and after chemotherapy.

II. To examine the relationship between blood estrogen levels and gut microbiota before and after chemotherapy.

TERTIARY OBJECTIVES:

I. To examine the relationship between changes in the gut microbiota by pre-treatment body mass index (BMI) (normal - BMI < 25 kg/m^2, overweight - BMI >= 25-< 30 kg/m^2, and obese- BMI >= 30 kg/m^2) and by changes in body composition in relation to chemotherapy.

OUTLINE: Patients are assigned to 1 of 3 groups.

GROUP A: Patients undergo collection of stool samples at baseline (before surgery), at 1 week before initiation of adjuvant chemotherapy (after surgery), and at 1 and 4 months after completion of adjuvant chemotherapy.

GROUP B: Patients undergo collection of stool samples at baseline (after surgery), at 1 week before initiation of adjuvant chemotherapy, and at 1 and 4 months after completion of adjuvant chemotherapy.

GROUP C: Patients undergo collection of stool samples at baseline, 1 month after completion of neoadjuvant chemotherapy (before surgery), and at 1 and 4 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ductal carcinoma in situ or invasive breast cancer (stage I, stage IIA, stage IIB, and stage IIIA breast cancer)
* A treatment group including surgery followed by standard treatment of adjuvant chemotherapy such as doxorubicin and cyclophosphamide followed by paclitaxel, docetaxel and cyclophosphamide, or a treatment group including neoadjuvant chemotherapy followed by surgery at the Norris or LAC+USC Medical Center
* Women of child-bearing potential agree to pregnancy test to confirm she is not pregnant
* Provide informed consent

Exclusion Criteria:

* Metastatic, recurrent, synchronous or metachronous breast cancer
* History of other cancers (other than non-melanoma skin cancer)
* History of autoimmune celiac or inflammatory bowel disease
* Past bariatric surgery
* Current or recent pregnancy or nursing (within past 12 months)
* Past treatment with chemotherapy
* Recent use (within past month) of more than 3 days of antibiotics use
* Current use of probiotic supplements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed breast cancer will be recruited from the Norris Comprehensive Cancer Center and the Los Angeles County + University of Southern California Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Change in intestinal microbiota (composition, abundance, and diversity) | Baseline to 4 months after final adjuvant (or neoadjuvant) chemotherapy course
  Paired sample t-test will be used to determine whether there are significant changes in microbiota diversity (as measured by the number of taxonomic groups) between pre-treatment levels and 1 and 4 months after the final chemotherapy treatment. Mixed-model linear regression on repeated measures will be used to concurrently adjust for physical activity, dietary intakes, and other factors.

SECONDARY OUTCOMES:
Change in body composition based on dual-energy x-ray absorptiometry (DEXA) | Baseline to 4 months after last chemotherapy
  Analyses of body composition measures will be based on fat mass, lean mass, and bone mineral content (BMC); each will be expressed in kilograms, on arms, legs, and trunk. Mixed effects regression models will be used to compare changes per week between pre-treatment assessment and 1 and 4 months after last chemotherapy. Additional analyses will use BMI group (normal, overweight, obese) for stratification and as a covariate in regression models. The relationship between body composition and gut microbiota before and after chemotherapy will be examined.
Baseline estradiol and estrone levels | Baseline
  Changes in the microbiota composition, abundance and diversity will be correlated with baseline estradiol and estrone levels.
Change in estrogen levels | Baseline to up to 4 months after last chemotherapy
  Correlation analyses of changes in the microbiota with changes in estrogen levels will be performed. Mixed effects regression analysis will be used to model systemic estrogen levels as a function of microbiota abundance and diversity, adjusting for cancer treatment, and baseline tumor and other individual characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wu, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States